CLINICAL TRIAL: NCT05626595
Title: PROmoting Early Childhood Outside (PRO-ECO) 2.0: A Program to Support Outdoor Play in Early Learning and Child Care Centres
Brief Title: PROmoting Early Childhood Outside 2.0
Acronym: PRO-ECO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Government of Canada (Other Government)
Responsible Party: Principal Investigator, Mariana Brussoni, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H20-01362
Record Dates: First submitted 2022-11-07; First posted 2022-11-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Child Development
Keywords: Children's outdoor play; Children's outdoor risky play; Early childhood education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Experimental): Outdoor play is an essential component of childhood development, including supporting children's cognitive, physical, emotional, and social growth. Currently, the early learning and childcare centres (ELCCs) host children within childcare settings, with outdoor playtime governed by institutional regulations.
  Interventions: Behavioral: Wait List Group - Normal Daily Practice
- Project (Sham Comparator): The PRO-ECO project to increase the quality of outdoor play involves four primary components:
  1. Modifying ELCC's outdoor play policies: the ELCC policy on outdoor play requirements and procedures will be modified in conjunction with ELCC management.
  2. ECE training and mentorship:
     ECEs will undergo the Learning Outside Together (LOT) program, which incorporates traditional wisdom into training on Indigenous ways of knowing, learning and experiencing the land as teacher.
  3. ELCC outdoor space modification:
     This includes designing and implementing tailored modifications for each centre's outdoor play space developed by landscape architecture students.
  4. Parent engagement:
  ELCCs will host parent-engagement events and opportunities to increase knowledge of the importance of outdoor play.
  Interventions: Behavioral: Project Group - PRO-ECO Project

INTERVENTIONS:
Behavioral: Project Group - PRO-ECO Project — The PRO-ECO project will be tailored to individual sites. Through collection of focus group and baseline data, the project will be further refined to provide site-specific adjustments, such as specific materials in the built environment design modification or targeted training. Identified features of effective projects outlined in the literature have informed the development of the project foundation and potential tailoring.
  Arms: Project
Behavioral: Wait List Group - Normal Daily Practice — ELCCs that are randomly assigned to the waitlist group will participate in their normal daily practice, including standard curriculum and outdoor play time. Once post-data collection is complete, wait list sites will be given the PRO-ECO project.
  Arms: Control

SUMMARY:
Licensed early learning and childcare centres (ELCCs) can provide children with rich opportunities for outdoor play that they may not otherwise experience in their home or community. However, many ELCCs struggle to provide high quality and stimulating outdoor play time. The primary aim of this study is to develop, implement and test a comprehensive multi-component project, the PROmoting Early Childhood Outside (PRO-ECO), to build capacity for, and address the complexities of building support for outdoor play in early childcare centre settings. This is to ultimately increase children's access to engaging outdoor spaces for play.

The overarching goal of this project is to develop and evaluate a comprehensive multi- component project, called the PROmoting Early Childhood Outside (PRO- ECO). This project is to increase children's outdoor play and the diversity of outdoor play behaviour in Canadian ELCC settings providing full-day licensed care for preschoolers. PRO-ECO integrates development of policies and procedure, early childhood educator (ECE) training and mentorship, outdoor space modifications and, parent/caregiver engagement.

The PRO-ECO project will be co-developed, implemented and evaluated in partnership with provincial childcare organizations and ten ELCCs. A wait-list control cluster randomised trial design (RCT) will evaluate the effectiveness of the project and how it can be modified to tackle barriers in diverse settings.

This project is an extension of the PRO-ECO pilot study (protocol ID H20-03912-A001, Clinicaltrials.gov ID NCT05073380).

DETAILED DESCRIPTION:
The design of this study is a wait-list control cluster randomised trial (RCT) with two arms. The two arms consist of 1) a PRO-ECO first project group and 2) a wait-list control group. The PRO-ECO project implementation consists of 4 primary components: 1) modifying existing/developing new ELCC policies and procedures related to outdoor play, 2) ECE training and mentorship through the Learning Outside Together program, providing outdoor play pedagogy theory and application, 3) ELCC outdoor space modification, and 4) parent and caregiver engagement of outdoor play activities.

A mixed-methods approach will be used to collect qualitative and quantitative data designed to meet the study objectives. Quantitative data collection will support evaluation of the primary outcome variables and qualitative data will be collected to assess the acceptability, effectiveness, and feasibility of the implementation of the project. Qualitative data will be collected concurrently with quantitative data and will allow researchers to explore how participants experience the project.

Participant inclusion and exclusion criteria are divided into three distinct sets of levels- 1) organization level, 2) adult individual participation, and 3) child participation.

1. Organization level Inclusion criteria of the ELCCs include approving participation in this study, readiness of the ELCC to participate and perceived need for the project (as assessed by the project partners and via interviews with the ELCCs). These variables will be measured based on a pretrial interview with ELCCs and key informants from the project steering committee. ELCCs that do not meet the inclusion characteristics based on these measurements may be excluded.
2. Adult individual participation Inclusion criteria for adult participants include being ECEs or staff (administrators, directors, and supervisors) at the participating ELCCs that provide full day childcare for preschool children.
3. Child individual participation Inclusion criteria for child participation includes being between the ages of 2.5-6 years, currently enrolled in one of the participating ELCCs, and obtaining parental consent for their participation in the study. Children will be excluded from the measurement portion of the study if their parent does not provide informed consent, however, all children attending the program will be exposed to the project.

The RCT will be conducted in 10 ELCCs across British Columbia. Individual ELCCs will serve as the unit of randomization, with 5 project sites and 5 wait-list control sites composing the final sample. Main project sites will receive the project deliverables immediately following baseline data collection, whereas wait-list control sites will receive the project deliverables 6 months later. Data on outcome measures will be collected at three time points: 1) Time 1 - Baseline, prior to project implementation, 2) Time 2 - 6-month follow-up (4 months following implementation of the project within the main project group, and 3) Time 3 - 12-month follow-up (10 months post-project for the main project group, 4 months post-intervention for the wait-list control group). Thus, outcome data will assess short-term and long-term outcomes within the project group and short-term outcomes within the wait-list control group. Baseline and post-project data will be included in the analysis, controlling for the cluster design.

Baseline and post-project data collection will occur during the Fall and Spring seasons to ensure similar weather patterns at all time points, which in British Columbia involves extensive rain and snow, depending on geographic area, as weather has been shown to impact outdoor play time.

As per study inclusion criteria, study participants will include children aged 2.5-6 years at 10 selected sites. This also includes the engagement of ECEs, supervisors, and managers. Parents of children will also be invited to participate in focus groups, consent provision, and information sharing. ELCCs will appoint a staff research lead to work closely with the research team on all phases of the project. Recruitment of children and parents will occur through the staff research lead at each ELCC. Letters and/or emails home and face-to- face conversations will promote recruitment. The research team will be actively involved with staff at each site to ensure they are provided information and direction on participant recruitment policies and procedures. The staff research lead at each ELCC will administer consent forms to families.

The investigators will inform parents/caregivers of children enrolled in the participating ELCCs about the study in various ways. This includes via online communications and info sessions. Adult participants for the qualitative focus group be recruited internally through the ELCC.

When contacted by prospective participants including ECEs and staff, the investigators will provide details of the study through phone, email or in-person connections. On the interview day, the consent and the overall interview procedure will be further explained to participants. The focus groups will be conducted through Zoom or in-person. Once procedures are explained and consent reviewed, the investigators will invite participants to sign the consent forms and complete the demographic survey, and email scanned copies to the UBC research team.

The outcome measures and methods for this study will be co-created with the project partners and may change after consultation. However, an overview of methods used within the pilot project that will guide this consultation are provided below.

For the primary outcome, children's time spent in bio play (engagement with natural environment elements) will be assessed utilizing observational behaviour mapping methods. To conduct observational behaviour mapping, two research staff will be on site at each of the 10 ELCCs to collect pre-determined data related to play behaviour during outdoor free play. Behaviour mapping assessments will be performed through scanning identified quadrants throughout the outdoor play space. Simultaneous to the in- situ coding, the project team, including research staff and ECE's, will be taking video recordings of the quadrants they are observing. Videos will be coded at 15-second intervals for play type, including bio play, physical play, expressive play, play with rules, imaginative play, exploratory play, restorative play, and non-play. Children's time spent in bio play will be calculated by adding up all measured/recorded time spent engaged in bio play. The investigators will compare time spent in bio play versus other play types at baseline and follow-up.

Children's participation in outdoor play will be assessed as a secondary outcome by comparing participation in play vs. non-play. Children's time spent in outdoor play will be calculated by adding up all measured/recorded time spent engaged in any type of play, excluding non-play. The diversity of children's play behavior when participating in outdoor play is also a secondary outcome and will be coded via observational behavior mapping methods. The investigators will compare the diversity of types of play occurring at baseline and follow- up by comparing proportions of the various play types, including physical play, expressive play, play with rules, imaginative play, exploratory play, restorative play, bio play, digital play and non-play.

ECEs' attitudes toward outdoor risky play is a secondary outcome and will be assessed using the Teacher Tolerance of Risk in Play Scale (T-TRiPS).

The quality of outdoor spaces will be an additional outcome. The Seven Cs audit tool will form the basis for the assessment of quality of outdoor space at all early childhood education centre sites, guide development of the plan for modification of the outdoor environment, and to reassess at main project early childhood education centre sites after implementation of the PRO-ECO project.

The same procedures described above will be followed to collect post- project data. The investigators will also collect ECEs and staff's acceptability of the PRO- ECO project. This will be done utilizing a combination of focus group discussion and administrative data.

ELIGIBILITY:
Participant inclusion and exclusion criteria is divided into three distinct sets of levels- 1) organization level, 2) adult individual participation, and 3) child participation.

1. The ELCC site inclusion criteria:

   We will select ELCCs providing full day care to preschool children to include in the study in consideration of readiness of program to participate and perceived need for the program, and time spent.
2. Adult participation inclusion criteria:

   Being early childhood educators (ECEs) or staff (e.g., administrators, directors and supervisors) at the participating ELCCs.
3. Child participation inclusion criteria:

   * Being between the ages of 2.5 to 6 years;
   * Currently enrolled in one of the participating ELCCs;
   * Obtained parental consent for their participation in the study.

Ages: 30 Months to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Assessing children's time spent in bio play | Project Group - Change of prevalence of bio play at 5-months and 10-months post-project implementation (Spring 2024 and Fall 2024); Wait List Control Group - Change of prevalence of bio play at 5-months post-project implementation (Fall 2024)
  To assess children's participation play that includes interaction with natural environment elements at ELCCs, an observational behavior mapping (OBM) methodology will be used. OBM involves understanding how an environment supports movement through mapping, recording, and analyzing geographically located data.

SECONDARY OUTCOMES:
Assessing the diversity of play types children engage in | Project Group - Change in play diversity at 5-months and 10-months post-project implementation (Spring 2024 and Fall 2024); Wait List Control Group - Change in play diversity at 5-months post-project implementation (Fall 2024)
  In addition to assessing time spent participating in outdoor free play, further detail on the type of play behaviour and movement is important to understanding children's outdoor free play in ELCC settings. OBM as described above will be used to assess the diversity of outdoor free play through 'play type'. Play types to be coded include physical play, expressive play, play with rules, imaginative play, exploratory play, restorative play, bio play, digital play and non-play.
Quality of early childhood education centres' outdoor play spaces | Project and Wait-list Control Group - Change in Seven C's Score at 5-months post-project implementation (Spring 2024; Fall 2024)
  The Seven Cs assessment tool, designed to provide guidance in the design of outdoor play spaces for children in early childhood settings, is based on seven criteria- character, context, connectivity, change, chance, clarity, and challenge. The Seven Cs will form the basis for the assessment and re-assessment of the quality of outdoor space at all centres, and will guide development of the plan for modification of the outdoor environment.
Early childhood educators' attitudes towards outdoor risky play | Project and Wait-list Control Group - Change in educators' attitudes at 5-months post-project implementation (Spring 2024; Fall 2024)
  The effect of the PRO-ECO project on early childhood educators' tolerance of risk in play will be assessed utilizing the Teacher Tolerance of Risk in Play Scale. The Teacher Tolerance of Risk in Play Scale is a 26-item yes/no survey question of risk tolerance; minimum = 0 and maximum = 26; higher scores mean a higher tolerance of risk in play.
Acceptability and feasibility of PRO-ECO project | Project and Wait-list Control Group - Change in educator and parent perspectives at 5-months post-project implementation (Spring 2024; Fall 2024)
  Qualitative data, including focus groups and/or individual key informant interviews, will be conducted with early childhood educators, early childhood education centre administrators, and parents respectively. Discussions will focus on how the project influenced the children and their outdoor play, as well as the groups' personal experiences with the project.
Assessing children's time spent in outdoor play | Project Group - Change of prevalence of play at 5-months and 10-months post-project implementation (Spring 2024 and Fall 2024); Wait List Control Group - Change of prevalence of play at 5-months post-project implementation (Fall 2024)
  To assess children's participation in outdoor free play at ELCCs, an observational behavior mapping (OBM) methodology will be used. OBM involves understanding how an environment supports movement through mapping, recording, and analyzing geographically located data.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Brussoni, Principal Investigator — University of British Columbia
Locations (10):
- Canada (10):
  - Curious Minds, Canal Flats, British Columbia
  - Outdoor Paradise, Cariboo, British Columbia
  - Turtle Island, Chetwynd, British Columbia
  - Kinnikinnick, Cranbrook, British Columbia
  - NW, Fort St. James, British Columbia
  - Ogopogo, Grand Forks, British Columbia
  - Bird's Nest, Lytton, British Columbia
  - Lily of the Valley, Surrey, British Columbia
  - The Nest, Victoria, British Columbia
  - Kulilu, Windermere, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
The data set will be available from Dr. Brussoni upon reasonable requests.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting upon publication of the RCT results until five years after publication.
Access Criteria: The data requests will be reviewed by the PRO-ECO Project Steering Committee, ELCC partners and Dr. Brussoni.

REFERENCES:
- [Derived] Brussoni M, Ramsden R, Grieve S, Mount D, Fox E, Herrington S, Lin Y, Johnson SE, Lloyd J, Elliot E, Mlieczko E, Lemire A, Scott L, Barrett A, Cottier E, Rice A. The 5 R's of Indigenous Research as a Framework to Co-Design and Evaluate an Outdoor Play Program in Early Learning and Child Care Centers: Protocol for the Promoting Early Childhood Outside (PRO-ECO) 2.0 Wait-List Control Cluster Randomized Trial. JMIR Res Protoc. 2025 Dec 12;14:e77956. doi: 10.2196/77956. PMID 41385788